CLINICAL TRIAL: NCT01108978
Title: Phase IV Study for Evaluating the Efficacy and Safety of Dehypotin® in the Patients With Type 2 Diabetes Mellitus or Cardiovascular Disease
Brief Title: Evaluating the Efficacy and Safety of Dehypotin® in the Patients With Type 2 Diabetes Mellitus or Cardiovascular Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Nang Kuang Pharmaceutical Co., Ltd. (Industry)
Collaborators: National Taiwan University Hospital (Other)
Responsible Party: Hsu Cindy, Nang Kuang Pharmaceutical Co., LTD
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 200911064M
Record Dates: First submitted 2010-04-21; First posted 2010-04-22 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2011-06

CONDITIONS: Type 2 Diabetes Mellitus; Cardiovascular Disease; Hypercholesterolemia
Keywords: Type 2 Diabetes Mellitus; Cardiovascular Disease; hypercholesterolemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Dehypotin (Active Comparator)
  Interventions: Drug: Dehypotin

INTERVENTIONS:
Drug: Placebo — Dehypotin® 40 mg/day or placebo, once a day, shortly after baseline for 12 consecutive weeks
  Arms: Placebo
Drug: Dehypotin — Dehypotin® 40 mg/day or placebo, once a day, shortly after baseline for 12 consecutive weeks
  Arms: Dehypotin

SUMMARY:
The purpose of this study is to evaluate the Efficacy and Safety of Dehypotin® in the Patients with Type 2 Diabetes Mellitus or Cardiovascular Disease. Eligible patients will be randomly assigned to 1 of 2 arms, either Dehypotin® or placebo, and will receive the diet advisement throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 20-75 years
* Diagnosis of type II Diabetes Mellitus for at least 3 months and/or clinical evident cardiovascular disease (CVD)
* A hemoglobin A1c concentration has to be < 8% before screening

Exclusion Criteria:

* Women of child bearing potential who are pregnant, breastfeeding or not using effective contraceptives
* Known hypersensitivity to Pravastatin or any of its components
* Have a history of homozygous familial hypercholesterolemia or known type III hyperlipoproteinemia
* Significant medical illness
* Known serious conditions, e.g. serum creatine kinase(CK)levels 2.5 times upper limit of normal
* Subjects being treated with drugs influence serum lipid concentrations
* Subjects who have cancer or been receiving the cancer chemotherapy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Evaluation absolute and percentage reductions in low-density lipoprotein cholesterol (LDL-C) by fasting biochemistry examination | 12-week treatment

SECONDARY OUTCOMES:
Evaluation of total cholesterol (TC), high-density lipoprotein cholesterol (HDL-C), triglycerides by fasting biochemistry examination | 12-week treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yang Wei Shiung, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Nang Kuang Pharmaceutical Co., LTD, Tainan, Xinhua Township, Taiwan